CLINICAL TRIAL: NCT04099342
Title: Enhanced Spatial Targeting in ECT Utilizing Focally Electrically-administered Seizure Therapy (FEAST)
Brief Title: Enhanced Spatial Targeting in ECT Utilizing FEAST
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: PI pausing to review clinical ECT and existing trials. Likely to resume.
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PSYCH-2019-27591
Record Dates: First submitted 2019-09-10; First posted 2019-09-23 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- A: FEAST (Experimental): Focally Electrically-administered Seizure Therapy (FEAST) is a form of Electroconvulsive therapy (ECT) that combines unidirectional stimulation, control of polarity, and an asymmetrical electrode configuration.
  Interventions: Device: FEAST; Device: FEAST RP
- B: RP FEAST (Experimental): Focally Electrically-administered Seizure Therapy (FEAST) with Reversed Polarity (RP) utilizes the same electrode placement as FEAST but a reversed directionality of current flow.
  Interventions: Device: FEAST; Device: FEAST RP

INTERVENTIONS:
Device: FEAST — FEAST with standard electrode configuration and current flow
Device: FEAST RP — FEAST with standard electrode configuration and reversed current flow

SUMMARY:
The purpose of this research study is to find an alternative version of ECT that reduces the negative side effects (mainly memory loss) while still providing patients with relief from depressive symptoms. Previous forms of ECT may use Bilateral (electrodes on both sides of the head) or Right Unilateral (RUL) (electrodes on one side of the head). Our research focuses on adjusting the placement of electrodes on one side of the head in order to better stimulate the Prefrontal Cortex (PFC) of the brain. By more specifically targeting the PFC, it is predicted that participants will receive the same benefit as ECT but will have fewer negative side effects after the treatment, mainly less memory loss. All other aspects of the treatment will be similar to regular, clinical ECT, including anesthesia and recovery monitoring. To accomplish this stimulation, an adjusted MECTA Spectrum 5000Q device will be used. If successful, this research study will demonstrate a way to improve ECT procedures for all patients suffering from Major Depressive Disorder by minimizing side effects and maintaining or improving efficacy.

DETAILED DESCRIPTION:
Study Design: This study will focus on refining FEAST methods by implementing a fixed-current titration and dosing method (800mA; 0.3 ms), testing the optimal directionality of current flow, and confirming specificity of induction of seizures in right orbitofrontal cortex. Twenty patients in an episode of major depression will be enrolled in the initial open-label study. Patients are kept on current medications for at least 2 weeks prior to initiation of therapy and throughout the treatment course. Patients are allowed PRN lorazepam limited to 3 mg/d but not within 10 hours of a FEAST session. Patients will undergo routine clinical care pre-ECT evaluations which include chemistry laboratory tests and an EKG. Patients will also undergo a brain MRI needed for 3D finite element modeling (FEM) to compute individual electric fields for each participant enrolled as well as an optional follow up MRI after treatment.

Once treatment is initiated, patients receive a dose 6 times initial Seizure Threshold (ST) at all treatments except the first and second, where ST is determined. If insufficient improvement (<40% change from baseline Hamilton Rating Scale for Depression, HRSD-24 item, or IDS-SR) after six treatments, the dose will increase by 50% in charge (9 times initial ST). Patients will undergo 6 channel EEG during all treatments. Participants will be randomized to FEAST (with typical electrodes placement and current flow directionality configurations) or Reverse Polarity FEAST to allow a direct comparison of induced seizure focality.

The primary measure right frontal to motor connectivity (seizure drive) and time for orientation recovery obtained following these sessions will permit direct comparison between normal configuration and RP FEAST as well. Preliminary data generated by the investigators suggest that RP polarity FEAST will elicit the most focal seizure with the shortest time for reorientation and fewest amnestic side effects.

Study Procedures:

A baseline appointment, scheduled at the Treatment Resistant Depression Clinic in Saint Louis Park, will be initially scheduled with potential participants to complete the informed consent process as well as baseline assessments for cognition, mood and quality of life. Participants will also undergo a baseline MRI that will consist of individual T1- and T2-weighted MRI scans which will be acquired with isotropic voxel resolution of 0.8 mm through resources located in the MIDB building. These structural data will be processed in the SimNIBS software to create a 3D volume conductor model of the subject's head. These MRI images will be constructed into 3D FEM models to compute non-invasive brain stimulation and electric fields for each participant enrolled.

All FEAST clinical procedures performed through Fairview will be documented in EPIC and duplicated in the research team's RedCap database for later analysis. Treatments are given in the morning, 3 times per week. Pharmacological agents are standardized: atropine (0.4 mg IV), methohexital (0.75 mg/kg) and succinylcholine (0.75-1.0 mg/kg). [If methohexital is unavailable, thiopental will be substituted (2.0 mg/kg]. Patients are oxygenated by mask (100% O2) prior to anesthesia and until resumption of spontaneous respiration. Standardized procedures are used to reduce impedance at ECT and EEG electrode sites. The d'Elia unilateral placement is used for conventional RUL ECT. FEAST will involve the 1.25" circular anterior electrode being centered at the measured FP2 position by the 10/20 EEG system, with the posterior cathode electrode (1"x2.5") tangential to the mid-sagittal plain and centered at vertex. FEAST is delivered with a modified MECTA Spectrum 5000Q relative to the commercial device with the capacity for unidirectional stimulation.

Follow up appointments after the 6th and 12th FEAST treatments (each within 1-2 days), as well as after the 15th session, if applicable, will also be conducted. They will include assessments of cognition, mood and quality of life. An optional follow up MRI may also be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of major depressive disorder using MINI-7 to derive RDC; DSM-IV
* Pretreatment HRSD score greater than or equal to 18
* ECT indicated by physician evaluation
* Willing and capable of providing informed consent as determined by physician evaluation

Exclusion Criteria:

* History of schizophrenia, schizoaffective disorder, other functional psychosis, or rapid cycling bipolar disorder as determined by MINI-7; rapid cycling defined as greater than or equal to four episodes in past year
* History of neurological illness or insult other than conditions associated with psychotropic exposure (e.g., tardive dyskinesia) determined by physician evaluation and medical history
* Alcohol or substance abuse or dependence in the past year (RDC) determined by physician evaluation
* Secondary diagnosis of a delirium, dementia, or amnestic disorder (DSM-IV), pregnancy, or epilepsy determined by physician evaluation
* Requires especially rapid antidepressant response due to suicidality, psychosis, inanition, psychosocial obligations, etc. determined by physician evaluation
* ECT in the past six months determined by physician evaluation and medical history
* Pregnancy as determined by urine pregnancy test and clinical interview

Ages: 22 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Seizure Drive Markers on EEG | 8 weeks
  Electrophysiological markers of the induced seizure will be captured with a 6-lead EEG placed over bilateral frontal, temporal and parietal lobes. Raw data will be collected in MicroVolts while the analysis will summarize connectivity measures. Right prefrontal activity and seizure drive will be contrasted to other regions from which EEG is recorded, to describe the focality of FEAST-induced seizures.
Seizure characteristics on EEG | 8 weeks
  Length of induced seizures is measured by EEG and recorded in seconds. Spectra powers, global and regional intensity will also be analyzed.
Seizure characteristics by motor observation | 8 weeks
  Length of induced seizures is measured by motor observation and recorded in seconds. Spectra powers, global and regional intensity will also be analyzed.

SECONDARY OUTCOMES:
Change in Hamilton Depression Rating Score (HDRS) | 8 weeks
  Change in HDRS from baseline to completion of each ECT treatment compared between 2 treatments - FEAST or FEAST RP. HDRS is a 24-item interview-based tool measuring depression symptoms in the previous week. Scoring is based on only the first 17 items. Eight items are scored on a 5-point scale, ranging from 0 = not present to 4 = severe. Nine are scored from 0-2. Total scores are the sum of the 17 item scores and range from 0 (Normal functioning) to 22 (severe depression).
Change in Inventory for Depressive Symptoms - Self Report (IDS-SR) Score | 8 weeks
  Change in IDS-SR scores from baseline to completion of each ECT treatment compared between 2 treatments - FEAST or FEAST RP. IDS-SR is a 30-item self report tool measuring depression symptoms in the previous week. Items are scored from 1 (normal functioning) to 3 (severely impaired) with some items scored on a yes (score of 1) or no (score of zero) basis. Items are summed to calculate the total score, which ranges from 0 (normal functioning) to 84 (severely impaired).
Time to Reorientation | 8 weeks
  Time between subject open eyes immediately after procedure and correctly identifying 4 out of 5 questions on orientation to name, time and space will be noted in seconds.
Amnestic Side Effects | 8 weeks
  Amnestic side effects will be determined via cognitive assessment and compared pre- and post-FEAST treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ziad Nahas, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States